CLINICAL TRIAL: NCT04317690
Title: Online Trial Examining Validity and Reliability of the Shared Decision Making Process Survey
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: University of Massachusetts, Boston (Other)
Responsible Party: Principal Investigator, Karen Sepucha, Director of the Health Decision Sciences Center, Massachusetts General Hospital
Other Study IDs: 2019P001434-1
Record Dates: First submitted 2020-03-19; First posted 2020-03-23 (Actual); Results first posted 2022-05-20 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: High Cholesterol; High Blood Pressure; Colorectal Cancer; Breast Cancer; Prostate Cancer
Keywords: shared decision making
MeSH Terms: conditions — Hypercholesterolemia; Hypertension; Colorectal Neoplasms; Breast Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- High Cholesterol: People between the ages of 30-75 ,with no previous heart attack or stroke history, who have been diagnosed with high cholesterol, who are either taking medication for high cholesterol for 2 years or less; or have discussed managing high cholesterol in the past 2 years. These people will see items only pertaining to high cholesterol.
- High Blood Pressure: People between the ages of 30-75 ,with no previous heart attack or stroke history, who have been diagnosed with high blood pressure, who are either taking medication for high blood pressure for 2 years or less; or have discussed managing high blood pressure in the past 2 years. These people will see items only pertaining to high blood pressure.
- Colorectal Cancer Screening: People between the ages of 50-75 with no previous diagnosis of colon cancer, who have been screened for colon cancer (or discussed screening for colon cancer) in the past 2 years, or who had first colon cancer screening in past 2 years. These people will see items only pertaining to colon cancer screening.
- Breast Cancer Screening: Females between the ages of 40-50 with no previous diagnosis of breast cancer who have had mammogram (or discussed having a mammogram) in the past 2 years, or had first mammogram in past 2 years. These people will see items only pertaining to breast cancer screening.
- Prostate Cancer Screening: Men between the ages of 45-69 with no previous diagnosis of prostate cancer who have been screened for prostate cancer (or discussed screening for prostate cancer) in the past 2 years or had first prostate cancer screening in the past 2 years. These people will see items only pertaining to prostate cancer screening.

SUMMARY:
The purpose of this study is to survey a sample of adults who have recently made a decision about treatment of high cholesterol or high blood pressure or a decision about screening for colorectal cancer, breast cancer, or prostate cancer. The main goal is to gather evidence of the validity and reliability of the Shared Decision Making Process scale. Secondary goal is to gather evidence on the quality of decisions for these common medical situations.

DETAILED DESCRIPTION:
Study staff worked with a national sampling firm to recruit subjects for five different medical decisions. The five decisions are (1) treatment of high cholesterol, (2) treatment of high blood pressure (3) when to start breast cancer screening (4) whether or not to have prostate cancer screening and (5) which test to have for colorectal cancer screening. Respondents complete a survey about their experiences talking with health care providers about the specific clinical decision. The survey measured the amount of shared decision making, knowledge, preferences, decisional conflict and decision regret. The study will obtain 500 responses total, or 100 for each decision.

Sample is an online non-probability panel of adults living in the United States. In the survey, participants were screened to meet specific qualifications. After 1 week, a random selection of 50 respondents are invited to complete the retest instrument.

All analyses will be conducted separately for each group, and results may be pooled across cancer screening and medication contexts. First, study staff will examine the descriptives for the Shared Decision Making Process items. Study staff will also test several hypotheses to examine validity of the scores such as whether higher shared decision making process scores are associated with less decisional conflict and less regret. Staff will also examine retest reliability of the Shared Decision Making Process scale.

ELIGIBILITY:
Inclusion Criteria:

High Blood Pressure Group

* Between the ages of 30-75
* No previous heart attack or stroke
* Have been diagnosed with high blood pressure
* Taking medication for high blood pressure for 2 years or less; or have discussed managing high blood pressure in the past 2 years

High Cholesterol

* Between the ages of 30-75
* No previous heart attack or stroke
* Have been diagnosed with high cholesterol
* Taking medication for high cholesterol for 2 years or less; or have discussed managing high cholesterol in the past 2 years

Colorectal Cancer Screening

* Between the ages of 50-75
* No previous diagnosis of colon cancer
* Have been screened for colon cancer (or discussed screening for colon cancer) in the past 2 years
* Had first colon cancer screening in past 2 years

Breast Cancer Screening

* Female
* Between the ages of 40-55
* No previous diagnosis of breast cancer
* Have had mammogram (or discussed having a mammogram) in the past 2 years
* Had first mammogram in past 2 years

Prostate Cancer Screening

* Male
* Between the ages of 45-69
* No previous diagnosis of prostate cancer
* Have been screened for prostate cancer (or discussed screening for prostate cancer) in the past 2 years
* Had first prostate cancer screening in past 2 years

Exclusion Criteria:

High Blood Pressure Group

* None

High Cholesterol

* None

Colorectal Cancer Screening

* None

Breast Cancer Screening

* None

Prostate Cancer Screening

* None

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sample was an online non-probability panel of adults living in the United States. Marketing Systems Group, the sample vendor, invited potential respondents from a targeted panel consisting of participants matching the sex, age, and group dynamics described above. In the survey, they were screened to meet our specific qualifications noted above.
Sampling Method: Non-Probability Sample
Enrollment: 539 (Actual)
Dates: Start 2020-03-17 (Actual); Primary Completion 2020-06-29 (Actual); Study Completion 2020-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Sepucha, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The study team will create a complete, cleaned, de-identified copy of the final data set for each online field test.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The data will be available t outside investigators starting 6 months after publication.
Access Criteria: Information about the data sets will be on the Health Decision Sciences Center website and in publications of the data. Dr. Sepucha will share a de-identified data set with outside investigators at no cost, according to approved Massachusetts General Hospital (MGH)/Partners policies for data sharing. Investigators from other sites will be able to request the data and will be required to complete a data use agreement that ensures that all local Institutional Review Board (IRB) requirements are met before using the data, that they will not attempt to identify any data in the dataset, and that they will not share the data set with anyone outside their project team.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: March 2020 - July 2020 using a national, non-probability panel obtained from Marketing Systems Group (MSG). MSG recruited participants by sending out invitation emails to potential responders.
Pre-assignment Details: Eligible respondents were adults in the US who had talked with a healthcare provider about screening for cancer (breast, colon, or prostate) or taking medication for a common chronic condition (depression, high cholesterol, or high blood pressure) in the past two years. Respondents were re-contacted approximately one-week post survey for a re-test survey.
Period: Overall Study
Arm/Group | High Cholesterol | High Blood Pressure | Colorectal Cancer Screening | Breast Cancer Screening | Prostate Cancer Screening
Started | 100 | 100 | 140 | 100 | 99
Completed | 100 | 96 | 140 | 98 | 99
Not Completed | 0 | 4 | 0 | 2 | 0
Not completed — did not have complete information for primary outcome | 0 | 4 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: participants who had discussed with their healthcare provider about cancer screening (breast, colon, prostate) or medication for a chronic condition (high cholesterol, high blood pressure) within the last 2 years. Participants needed to have provided enough information to calculate the shared decision making process score (primary outcome of interest)
Groups:
- Total: Total of all reporting groups
Arm/Group | High Cholesterol | High Blood Pressure | Colorectal Cancer Screening | Breast Cancer Screening | Prostate Cancer Screening | Total
Number analyzed (Participants) | 100 | 96 | 140 | 98 | 99 | 533
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (12) | 43 (11) | 61 (7) | 44 (3) | 52 (4) | 52 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 41 | 43 | 98 | 0 | 245
  Male | 37 | 55 | 97 | 0 | 99 | 288
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 11 | 10 | 8 | 6 | 45
  Not Hispanic or Latino | 90 | 85 | 130 | 90 | 93 | 488
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 0 | 1 | 3
  Asian | 4 | 2 | 4 | 7 | 0 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 8 | 11 | 16 | 9 | 17 | 61
  White | 78 | 74 | 112 | 75 | 75 | 414
  More than one race | 3 | 4 | 2 | 2 | 1 | 12
  Unknown or Not Reported | 7 | 4 | 5 | 5 | 5 | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Shared Decision Making Process Measure
Description: The Shared Decision Making Process is a short patient-reported survey that measures the amount of shared decision making that occurs in an interaction. Scores range from 0-4 where higher values indicate a better shared decision making process occurred.
Time Frame: Baseline survey
Population: participants who provided complete information to calculate a shared decision making process score (primary outcome of interest)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Cholesterol | High Blood Pressure | Colorectal Cancer Screening | Breast Cancer Screening | Prostate Cancer Screening
Number analyzed (Participants) | 100 | 96 | 140 | 98 | 99
score on a scale | 2.12 (1.03) | 2.65 (1.04) | 1.61 (1.12) | 1.4 (1.1) | 1.87 (0.97)

2. Secondary Outcome: Decisional Conflict Tool (SURE)
Description: Measures decisional conflict, consists of 4 yes/no items. Scores range 0-4 where 0 indicates no decisional conflict, and scores 1 to 3 indicate decisional conflict. The measure is often reported as a top-score of 0, thus the percentage of patients with a total score of 0 or no decisional conflict.
Time Frame: Baseline survey
Population: participants who completed all 4 items of the short decisional conflict scale. Only 532/533 participants provided enough information to calculate a SURE score.
Measure: Number; unit: percentage of participants
Arm/Group | High Cholesterol | High Blood Pressure | Colorectal Cancer Screening | Breast Cancer Screening | Prostate Cancer Screening
Number analyzed (Participants) | 100 | 96 | 139 | 98 | 99
percentage of participants | 68 | 70 | 68 | 78 | 71

3. Secondary Outcome: Decision Regret Scale
Description: 5-item decision regret scale ranges from 0-100 with higher scores indicating greater decisional regret.
Time Frame: Baseline survey
Population: Participants who answered all 5 decision regret questions. Only 526/533 participants provided enough information to calculate decision regret score.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Cholesterol | High Blood Pressure | Colorectal Cancer Screening | Breast Cancer Screening | Prostate Cancer Screening
Number analyzed (Participants) | 100 | 94 | 139 | 95 | 98
score on a scale | 22 (18) | 27 (18) | 17 (18) | 16 (16) | 25 (22)

4. Secondary Outcome: Single-Item Measure of Decision Regret
Description: Single item asking "If you knew then what you know now, do you think you would make the same decision about [how to manage your high cholesterol/ how to manage your high blood pressure/breast cancer screening/colon cancer screening/ prostate cancer screening]?" where the last part varies by group.
  Response options are:
  Definitely yes, Probably yes, Probably no, Definitely no
Time Frame: Baseline survey
Population: participants who answered the single-item regret question.
Measure: Count of Participants; unit: Participants
Arm/Group | High Cholesterol | High Blood Pressure | Colorectal Cancer Screening | Breast Cancer Screening | Prostate Cancer Screening
Number analyzed (Participants) | 100 | 96 | 140 | 98 | 99
Participants
  Definitely yes | 49 | 52 | 77 | 61 | 50
  Probably yes | 44 | 37 | 54 | 32 | 39
  Probably no | 5 | 7 | 8 | 4 | 7
  Definitely no | 2 | 0 | 1 | 1 | 3

5. Secondary Outcome: Treatment Choice
Description: Single item asking patient "What did you want to do" in regard to (depending on the group) high cholesterol/high blood pressure/colon cancer screening/breast cancer screening/prostate cancer screening
Time Frame: Baseline survey
Population: participants who answered the treatment preference question.
Measure: Count of Participants; unit: Participants
Arm/Group | High Cholesterol | High Blood Pressure | Colorectal Cancer Screening | Breast Cancer Screening | Prostate Cancer Screening
Number analyzed (Participants) | 100 | 96 | 140 | 97 | 99
Participants
  take medicine/(start) screen for cancer | 37 | 64 | 123 | 72 | 71
  not take medicine/(wait) not screen for cancer | 61 | 32 | 16 | 19 | 25
  other | 2 | 0 | 1 | 6 | 3

6. Secondary Outcome: Adapted Controlled Preference Scale
Description: Single item asking the participant who made the ultimate decision. The categorical response options are 1) the patient made the decision, 2)the provider made the decision, or 3) both patient and provider made the decision together.
Time Frame: Baseline survey
Population: participants who answered the controlled preference scale question.
Measure: Count of Participants; unit: Participants
Arm/Group | High Cholesterol | High Blood Pressure | Colorectal Cancer Screening | Breast Cancer Screening | Prostate Cancer Screening
Number analyzed (Participants) | 100 | 96 | 140 | 98 | 99
Participants
  Mainly my decision | 43 | 46 | 59 | 49 | 68
  Mainly the healthcare provider's decision | 18 | 24 | 25 | 13 | 10
  We made the decision together | 39 | 26 | 56 | 36 | 21

7. Secondary Outcome: Shared Decision Making Process Measure Retest
Description: as for outcome 1
Time Frame: 1 week after baseline survey
Population: Participants who completed the baseline survey were re-contacted approximately 1 week post-survey for a retest. Participants who completed the retest survey and provided enough information to calculate the shared decision making process score were part of this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Cholesterol | High Blood Pressure | Colorectal Cancer Screening | Breast Cancer Screening | Prostate Cancer Screening
Number analyzed (Participants) | 45 | 40 | 65 | 42 | 38
score on a scale | 2.27 (1.02) | 2.32 (1.42) | 1.68 (1.13) | 1.57 (1.18) | 1.67 (1.02)

8. Secondary Outcome: Knowledge
Description: Multiple choice knowledge items for each topic will be combined to a total knowledge score (0-100) with higher scores indicating higher knowledge
Time Frame: Baseline survey
Population: participants who answered at least 50% of the knowledge items in their respective clinical groups. Participants in the high cholesterol group were not given a knowledge score. Only 131/234 provided enough information to calculate a shared decision making process score (primary outcome of interest)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Cholesterol | High Blood Pressure | Colorectal Cancer Screening | Breast Cancer Screening | Prostate Cancer Screening
Number analyzed (Participants) | 0 | 96 | 137 | 98 | 99
score on a scale |  | 61 (29) | 56 (22) | 40 (18) | 43 (26)

9. Other Pre Specified Outcome: Adherence
Description: 3 item measure of adherence to medication asked for the high cholesterol and high blood pressure sample participants who indicate that they are taking medicine. (patients in the cancer screening arm did not get this question). composite score ranged from 0-100, with higher scores indicating greater adherence to medication within the last 30 days.
Time Frame: Baseline survey
Population: participants in the high cholesterol and high blood pressure groups who answered all 3 medication adherence questions. participants in the three cancer screening groups were not assigned medication adherence questions and thus were not part of this analysis. Only 56/100 (high cholesterol) and 68/96 (high blood pressure) participants provided enough information to calculate adherence score.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Cholesterol | High Blood Pressure | Colorectal Cancer Screening | Breast Cancer Screening | Prostate Cancer Screening
Number analyzed (Participants) | 56 | 68 | 0 | 0 | 0
score on a scale | 85 (19) | 87 (14) |  |  |

ADVERSE EVENTS:
Time Frame: Surveys responses were reviewed within 2 weeks of completion for evidence of adverse events
Description: Our definition of adverse event and/or serious adverse event did not differ.
Arm/Group | High Cholesterol | High Blood Pressure | Colorectal Cancer Screening | Breast Cancer Screening | Prostate Cancer Screening
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/100 | 0/140 | 0/100 | 0/99
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/100 | 0/140 | 0/100 | 0/99
Other Adverse Events (participants affected / at risk) | 0/100 | 0/100 | 0/140 | 0/100 | 0/99

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-18): https://cdn.clinicaltrials.gov/large-docs/90/NCT04317690/Prot_SAP_000.pdf